CLINICAL TRIAL: NCT02238925
Title: An Open Label Phase II Pharmacokinetic and Pharmacodynamic Assessment of the Potential for QTc Prolongation Following First Induction Treatment With CPX-351 (Cytarabine:Daunorubicin) Liposome Injection in Acute Leukemias and MDS Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTR0310-206
Record Dates: First submitted 2014-08-14; First posted 2014-09-12 (Estimated); Results first posted 2017-11-30 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-10

CONDITIONS: Acute Myeloid Leukemia (AML); Acute Lymphoblastic Leukemia (ALL); Myelodysplastic Syndrome (MDS)
Keywords: Newly Diagnosed AML; Secondary AML; Relapsed/Refractory AML; Relapsed/Refractory ALL; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Recurrence | interventions — CPX-351

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CPX-351 (Experimental): Single Arm Study (Patients may receive up to 2 Inductions and 4 Consolidations):
  Induction 1: CPX-351 will be given intravenously at 100units/m2 on days 1, 3, and 5 over a 90 minute infusion.
  Induction 2: CPX-351 will be given intravenously at 100units/m2 on days 1 and 3 over a 90 minute infusion.
  Consolidations 1-4: CPX-351 will be given intravenously at 65units/m2 on days 1 and 3 over a 90 minute infusion.
  Interventions: Drug: CPX-351

INTERVENTIONS:
Drug: CPX-351

SUMMARY:
The purpose of this study is to assess the effects of CPX-351 on cardiac repolarization, assess plasma drug levels, asses serum copper levels, and assess drug levels in urine.

Efficacy and Safety will be assessed in all patients enrolled to the study.

DETAILED DESCRIPTION:
This study is an open-label, single-arm, Phase II, PK and pharmacodynamic (PD) trial of CPX-351 in patients with documented acute leukemia (AML or ALL) or MDS (IPSS score ≥ 1.5) and suitable for treatment with intensive chemotherapy. Each patient will be screened for hepatic impairment. Hepatic impairment will be assessed using the Child-Pugh system and only patients with a Child-Pugh score <7 points will be eligible for this study. Patients will receive up to two inductions and four consolidation courses. Patients will be monitored for safety (early deaths, adverse events, metabolic changes, etc.) and efficacy (response for AML, ALL, and MDS) while on the study.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and voluntarily sign an informed consent form
* Age ≥ 18 to ≤ 80 years at the time of signing the informed consent form
* Life expectancy of at least 3 months
* Pathological confirmation by bone marrow documenting the following:

  * Newly Diagnosed De novo AML according to WHO criteria except for Acute Promyelocytic Leukemia or patients with known favorable cytogenetics (see exclusion)
  * Newly Diagnosed Secondary AML age <60 years and ≥76 to 80 years, defined as having a history of an antecedent hematologic disorder (myelodysplastic syndromes [MDS], myeloproliferative disease [MPD]or history of cytotoxic treatment for non-hematologic malignancy)
  * Patients with relapsed/refractory AML regardless of cytogenetic risk
  * Patients with relapsed/refractory ALL
  * Patients with MDS (IPSS score ≥ 1.5)
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0-2
* Able to adhere to the study visit schedule and other protocol requirements
* Laboratory values fulfilling the following:

  * Serum Creatinine ≤ 2.0mg/dL
  * Hepatic function with a score of < 7 points according to the Child-Pugh System
  * Serum alanine aminotransferase or aspartate aminotransferase < 3 times the ULN. Note: If elevated liver enzymes are related to disease; contact medical monitor to discuss.
* Cardiac ejection fraction ≥50% by ECHO or MUGA
* Screening and Baseline QTcF (Fridericia's) less than 470 msec
* Patients with second malignancies in remission may be eligible if there is clinical evidence of disease stability for a period of greater than 6 months off cytotoxic chemotherapy, documented by imaging, tumor marker studies, etc., at screening. Patients maintained on long-term non-chemotherapy treatment, e.g., hormonal therapy, are eligible.
* All men and women must agree to practice effective contraception during the study period if not otherwise documented to be infertile.

Exclusion Criteria:

* Patients eligible for participation in Study CLTR0310-301 (Phase III study of CPX-351 NCT01696084) or who have already participated in that study are not eligible for this study.
* Patients taking medications known to prolong the QTc interval directly or that interact pharmacodynamically with medicines to prolong the QTc interval.
* Rhythm abnormalities (other than sinus bradycardia with HR < 50 bpm)
* AV block (other than 1o AV Block with PR > 200 msec)
* Bundle branch block or QRS ≥ 120 msec
* Abnormal T wave morphology (other than slight flattening)
* Pathological U waves
* Other QRS or T/U morphology preventing accurate determination of QT interval
* Patients with unexplained syncope, history of or known risk factors for torsade des pointes, including congenital long QT syndrome, or family history of LQTS.
* Patients with history of and/or current evidence of myocardial impairment (e.g. cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (Class III or IV staging)
* Newly diagnosed patients with Acute promyelocytic leukemia [t(15;17)] or favorable cytogenetics, including t(8;21) or inv16
* Clinical evidence of active CNS leukemic involvement
* Chemotherapy or other investigational anticancer therapeutic drugs within 1 week prior to study entry unless AEs have resolved and there is no interference with the assessment of efficacy or safety; in the event of rapidly proliferative disease, however, the use of hydroxyurea is permitted up to 12 hours before study entry. Patients with prior bone marrow or stem cell transplant, considered for inclusion, should be discussed with the medical monitor first.
* Any serious medical condition or psychiatric illness that would prevent the patient from providing informed consent
* Patients with prior cumulative anthracycline exposure of greater than 368 mg/m2 daunorubicin (or equivalent)
* Active or uncontrolled infection. Patients with any infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for ≥72 hrs. Patients with fevers believed to be due to leukemia or MDS are eligible provided a thorough infection work-up is negative and the patient is clinically and hemodynamically stable.
* Pregnant or lactating women
* Hypersensitivity to cytarabine, daunorubicin or liposomal products
* History of Wilson's disease or other copper-related metabolic disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-07; Primary Completion 2015-05 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Franciscan Saint Francis Health, Indianapolis, Indiana
  - University of Kansas Cancer Center, Westwood, Kansas
  - Oregon Health & Science University, Portland, Oregon
  - Medical University of South Carolina, Charleston, South Carolina
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Lin TL, Newell LF, Stuart RK, Michaelis LC, Rubenstein E, Pentikis HS, Callahan T, Alvarez D, Liboiron BD, Mayer LD, Wang Q, Banerjee K, Louie AC. A phase 2 study to assess the pharmacokinetics and pharmacodynamics of CPX-351 and its effects on cardiac repolarization in patients with acute leukemias. Cancer Chemother Pharmacol. 2019 Jul;84(1):163-173. doi: 10.1007/s00280-019-03856-9. Epub 2019 May 16. PMID 31098682

RESULTS

PARTICIPANT FLOW:
Groups:
- CPX-351: Single Arm Study (Patients may receive up to 2 Inductions and up to 4 Consolidations):
  Induction 1: CPX-351 will be given intravenously at 100units/m2 on days 1, 3, and 5 over a 90 minute infusion.
  Induction 2: CPX-351 will be given intravenously at 100units/m2 on days 1 and 3 over a 90 minute infusion.
  Consolidations: CPX-351 will be given intravenously at 65units/m2 on days 1 and 3 over a 90 minute infusion.
  CPX-351
Period: Overall Study
Arm/Group | CPX-351
Started | 26
Completed | 1
Not Completed | 25

BASELINE CHARACTERISTICS:
Arm/Group | CPX-351
Number analyzed (Participants) | 26
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (9.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 14

OUTCOME MEASURES:

1. Primary Outcome: Effect of CPX-351 on Cardiac Ventricular Repolarization (QTcF)
Description: Time-matched QTcF Changes From Baseline after the start of first infusion
Time Frame: 21 days
Population: All subjects who received any dose of study drug and had at least 1 time-matched change from baseline in ECG parameters.
Measure: Mean (Standard Deviation); unit: msecs
Arm/Group | CPX-351
Number analyzed (Participants) | 26
msecs
  Time-point 0.75 h | 0.6 (15.13)
  Time-point 1.5 h | -1.2 (13.30)
  Time-point 2 h | 4.3 (15.96)
  Time-point 3 h | 5.3 (15.17)
  Time-point 4 h | 8.0 (11.69)
  Time-point 6 h | -0.1 (11.24)
  Time-point 8 h | 4.8 (8.52)
  Time-point 12 h | -2.3 (10.43)
  Time-point 24 h | -6.2 (13.91)

2. Secondary Outcome: Serum Copper Levels Change From Baseline
Description: Change from Baseline to Induction 1, Day 5
Time Frame: During 1st induction (up to 5 days)
Population: All subjects who received at least 1 dose of study drug and copper data were collected.
Measure: Mean (Standard Deviation); unit: μg/dL
Arm/Group | CPX-351
Number analyzed (Participants) | 24
μg/dL | 64.95 (51.119)

3. Secondary Outcome: Complete Response Rate
Time Frame: Following 1st induction, following 2nd induction if applicable
Population: Efficacy population: All subjects who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | CPX-351
Number analyzed (Participants) | 26
Participants | 8

4. Secondary Outcome: Tmax
Time Frame: Induction 1, Day 5
Measure: Median (Full Range); unit: hours
Arm/Group | CPX-351
Number analyzed (Participants) | 26
hours
  Cytarabine | 2.00 [0.75 to 8.33]
  Ara-U | 8.00 [5.78 to 8.33]
  Daunorubicin | 2.00 [0.75 to 6.02]
  Daunorubicinol | 26.00 [1.50 to 48.00]

5. Secondary Outcome: Cmax
Time Frame: Induction 1, Day 5
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | CPX-351
Number analyzed (Participants) | 26
ng/ml
  Cytarabine | 62200 (20900)
  Ara-U | 1240 (252)
  Daunorubicin | 26000 (8510)
  Daunorubicinol | 147 (52.3)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the start of infusion to the last day of the study period, whereas Serious Adverse Events were reported from the start of infusion until 30 days after completion of the study period.
Description: The Safety population included subjects receiving at least 1 dose of study drug.
Arm/Group | CPX-351
Serious Adverse Events (participants affected / at risk) | 8/26
Other Adverse Events (participants affected / at risk) | 26/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-351 (N=26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 7
Ileus (Gastrointestinal disorders) | 1
Catheter Site Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Meningitis Bacterial (Infections and infestations) | 1
Pathogen Resistance (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pulmonary Mycosis (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Ejection Fraction Decreased (Investigations) | 1
Acute Myeloid Leukamia Recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CPX-351 (N=26)
Febrile Neutropenia (Blood and lymphatic system disorders) | 17
Sinus Tachycardia (Cardiac disorders) | 5
Tachycardia (Cardiac disorders) | 4
Blepharospasm (Eye disorders) | 2
Conjunctival Haemorrhage (Eye disorders) | 2
Dry Eye (Eye disorders) | 2
Vitreous Floaters (Eye disorders) | 2
Nausea (Gastrointestinal disorders) | 14
Diarrhoea (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 11
Vomiting (Gastrointestinal disorders) | 10
Abdominal Pain (Gastrointestinal disorders) | 6
Gingival Bleeding (Gastrointestinal disorders) | 4
Abdominal Pain Lower (Gastrointestinal disorders) | 3
Dysphagia (Gastrointestinal disorders) | 3
Faecal Incontinence (Gastrointestinal disorders) | 3
Stomatitis (Gastrointestinal disorders) | 3
Cheilitis (Gastrointestinal disorders) | 2
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2
Gingival Pain (Gastrointestinal disorders) | 2
Haemorrhoids (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 14
Oedema Peripheral (General disorders) | 10
Chills (General disorders) | 7
Pyrexia (General disorders) | 6
Gait Disturbance (General disorders) | 3
Mucosal Inflammation (General disorders) | 3
Non-Cardiac Chest Pain (General disorders) | 3
Nodule (General disorders) | 2
Bacteraemia (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Cellulitis (Infections and infestations) | 2
Clostridium Difficile Colitis (Infections and infestations) | 2
Device Related Infection (Infections and infestations) | 2
Folliculitis (Infections and infestations) | 2
Staphylococcal Bacteraemia (Infections and infestations) | 2
Contusion (Injury, poisoning and procedural complications) | 3
Excoriation (Injury, poisoning and procedural complications) | 2
Human Rhinovirus Test Positive (Investigations) | 2
Viral Test Positive (Investigations) | 2
Weight Decreased (Investigations) | 2
Weight Increased (Investigations) | 2
Decreased Appetite (Metabolism and nutrition disorders) | 12
Fluid Overload (Metabolism and nutrition disorders) | 3
Fluid Retention (Metabolism and nutrition disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 6
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Neck Pain (Musculoskeletal and connective tissue disorders) | 5
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 3
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 3
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 2
Headache (Nervous system disorders) | 11
Dizziness (Nervous system disorders) | 5
Dizziness Postural (Nervous system disorders) | 3
Tremor (Nervous system disorders) | 3
Ataxia (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Sinus Headache (Nervous system disorders) | 2
Insomnia (Psychiatric disorders) | 11
Confusional State (Psychiatric disorders) | 6
Depression (Psychiatric disorders) | 4
Agitation (Psychiatric disorders) | 3
Anxiety (Psychiatric disorders) | 2
Delirium (Psychiatric disorders) | 2
Sleep Disorder (Psychiatric disorders) | 2
Chromaturia (Renal and urinary disorders) | 4
Pollakiuria (Renal and urinary disorders) | 4
Urinary Incontinence (Renal and urinary disorders) | 4
Haematuria (Renal and urinary disorders) | 3
Dysuria (Renal and urinary disorders) | 2
Micturition Urgency (Renal and urinary disorders) | 2
Urinary Retention (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 7
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3
Rales (Respiratory, thoracic and mediastinal disorders) | 3
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary Mass (Respiratory, thoracic and mediastinal disorders) | 2
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Upper-Airway Cough Syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 5
Erythema (Skin and subcutaneous tissue disorders) | 4
Petechiae (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3
Rash Erythematous (Skin and subcutaneous tissue disorders) | 3
Rash Papular (Skin and subcutaneous tissue disorders) | 3
Rash Pruritic (Skin and subcutaneous tissue disorders) | 3
Blood Blister (Skin and subcutaneous tissue disorders) | 2
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 2
Purpura (Skin and subcutaneous tissue disorders) | 2
Rash Macular (Skin and subcutaneous tissue disorders) | 2
Skin Mass (Skin and subcutaneous tissue disorders) | 2
Hypotension (Vascular disorders) | 8
Hypertension (Vascular disorders) | 4
Flushing (Vascular disorders) | 2
Haematoma (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No